CLINICAL TRIAL: NCT04017728
Title: Percutaneous Vertebroplasty Using Rotary Cutter for Treating Bone Metastases
Brief Title: Percutaneous Vertebroplasty Using Rotary Cutter for Bone Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 960HP20190051
Record Dates: First submitted 2019-04-13; First posted 2019-07-12 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Percutaneous Vertebroplasty (Active Comparator): The cement is injected after the successful puncture.
  Interventions: Device: Conventional Percutaneous Vertebroplasty
- Percutaneous Vertebroplasty with Rotary Cutter (Experimental): The rotary cutter is applied to destroy the metastatic lesion before coment injection.
  Interventions: Device: Percutaneous Vertebroplasty with Rotary Cutter

INTERVENTIONS:
Device: Conventional Percutaneous Vertebroplasty — The cement is injected into the bone metastases directly.
  Arms: Conventional Percutaneous Vertebroplasty
Device: Percutaneous Vertebroplasty with Rotary Cutter — The rotary cutter is applied before the cement injection. Then, the cement is injected with lower pressure.
  Arms: Percutaneous Vertebroplasty with Rotary Cutter

SUMMARY:
Percutaneous vertebroplasty has been applied widely to treat bone metastases. The injected cement may strengthen the affected bone to prevent pathological fractures and relieve the pain. Moreover, the thermal reaction (70°C) due to polymerisation of cement also contributes to tumour destruction. The cement dose and diffusion pattern may be significant factors for the treatment efficacy, which can be affected by the inner pressure of the metastases. The investigators will apply a rotary cutter to destroy the structure of metastases to alleviate the pressure in the metastases. Then, more cement will be injected, which may effectively interdigitates with the surrounding bone and generate more thermo to kill the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging-proven and pathology-proven metastases
2. Intractable pain with neurologic dysfunction

Exclusion Criteria:

1. Poor general condition without tolerance of surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-07-30 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Back pain: Visual analogue scales system | 3 months
  Measuring and comparing the pre- and post-operative back pain via Visual analogue scales (VAS) system with values from 0 to 10 (0 indicating no pain and 10 indicating the worst pain). Patients with a VAS score lower than 3 were classified as the effective group.

SECONDARY OUTCOMES:
The patterns of cement opacification | during the procedure of vertebroplasty
  The patterns of cement opacification were classified as solid patterns (cement forms a mass), trabecular patterns (cement spread along the fine bone trabeculae), and mixed patterns (cement forms a mass with spreading along the fine bone trabeculae).
Cement leakage | during the procedure of vertebroplasty
  The presence or absence of cement leakage is assessed in the groups with and without rotary cutter.
Cement volume | during the procedure of vertebroplasty
  The injected cement volume were evaluated in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- 960 Hospital of PLA, Jinan, Shandong, China